CLINICAL TRIAL: NCT06309823
Title: A Single-patient Clinical Trial of MAS825 in a Patient With XIAP Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dilan Dissanayake, Project Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000080330
Record Dates: First submitted 2024-02-23; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: X-linked Lymphoproliferative Syndrome Type 2 (XLP-2)
MeSH Terms: conditions — Lymphoproliferative Syndrome, X-Linked, 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Active treatment (Experimental)
  Interventions: Drug: MAS825

INTERVENTIONS:
Drug: MAS825 — MAS825 is a bi-specific IgG1 monoclonal antibody that simultaneously targets IL-1beta and IL-18, thereby neutralizing both cytokines that are thought to be integral to the pathogenesis of XLP-2.

SUMMARY:
MAS825 is a bi-specific IgG1 monoclonal antibody that simultaneously targets IL-1 beta and IL-18, thereby neutralizing both cytokines that are thought to be integral to the pathogenesis of XLP-2. Clinical trials are currently examining its efficacy in other diseases associated with elevations of these cytokines, including NLRC4-associated disease and hidradenitis suppurativa. This study proposes to assess the effectiveness of MAS825 in a single patient with XLP-2, who has previously demonstrated response to blockade of IL-1 beta and IL-18. Given the lack of alternative pharmaceutical options for XLP-2, this represents the only known medication option that avoids the toxicity associated with high-dose corticosteroids and the morbidity associated with hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Known patient with XIAP genetic defect under the care of the investigator

Exclusion Criteria:

* N/A

Ages: 13 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Impact of MAS825 on Physician Global Assessment Score | 5 years
  Likert Scale:
  0 = Absent (no) disease associated clinical signs and symptoms
  1. = Minimal disease associated signs and symptoms
  2. = Mild disease associated signs and symptoms
  3. = Moderate disease associated signs and symptoms
  4. = Severe disease associated signs and symptoms
Impact of MAS825 on Physician Severity Assessment of Disease Signs and Symptoms | 5 years
  The signs and symptoms assessed include: 1) Abdominal pain 2) Diarrhea 3) Fever using a Likert scale:
  0 = Absent
  1. = Minimal
  2. = Mild
  3. = Moderate
  4. = Severe
Patient/Parent Global Assessment of Disease Activity | 5 years
  Likert Scale:
  0 = Absent (no) disease associated clinical signs and symptoms
  1. = Minimal disease associated signs and symptoms
  2. = Mild disease associated signs and symptoms
  3. = Moderate disease associated signs and symptoms
  4. = Severe disease associated signs and symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada